CLINICAL TRIAL: NCT05159362
Title: Reward-based Technology to Improve Opioid Use Disorder Treatment Initiation After an ED Visit - Phase 1
Brief Title: Usability Testing for the Reward-based Technology to Improve OUD Treatment
Acronym: OARSCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Q2i, LLC (Industry)
Collaborators: University of Massachusetts, Worcester (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H00017879-1; R42DA049448 (NIH)
Record Dates: First submitted 2021-10-20; First posted 2021-12-16 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Opioid-use Disorder; Contingency Management; Medication for Opioid-use Disorder
Keywords: Substance Use Disorder; Opioid Use Disorder; Contingency Management; Medication for opioid use disorder; Medication-assisted treatment
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants were enrolled and monitored through a 4-week field test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OARSCM (Experimental): After successful completion of usability testing (Patients: n=12, Providers: n=4), a proof-of-concept field test was completed. OARSCM patients (n = 11) received TAU procedures during enrollment (SBIRT for opioid use disorder and a warm handoff to outpatient MOUD treatment). TAU outpatient MOUD treatment consists of urine toxicology (Utox) screening, group/individual therapy, and MOUD prescription. Treatment visits are typically weekly in weeks 1-4 and taper over time. Patients earned chances for prizes, for targeted behaviors, which escalated for each targeted behavior in a row, with reset criteria. For scheduling a MOUD treatment intake, patients will earn 2 chances for prizes. Chances for prizes will increase by 2 chances with each targeted behavior in a row up to a max of 10 draws/targeted behavior. There are 18 targeted behaviors during the 4-week field test (schedule intake, complete intake, 4 opioid-negative Utox/week plus bonuses for cocaine-negative Utox, and 4 therapy/week).
  Interventions: Other: Software Application

INTERVENTIONS:
Other: Software Application — Access is granted to participants for 4 weeks to the OARSCM platform which includes reinforcements for meeting MOUD treatment goals.
  Other Names: Opioid Addiction Recovery Support - Contingency Management (OARSCM)

SUMMARY:
Millions of people in the US misuse opioids each year, leading to thousands of deaths and costing billions of dollars in total economic burden. Medication assisted treatment (MAT) for opioid use disorder (OUD) is highly efficacious, but only a fraction of OUD persons access MAT, and treatment non-adherence is common and associated with poor outcomes. This STTR Fast Track proposal is designed to increase rates of Suboxone (buprenorphine/naloxone) treatment initiation and adherence among OUD patients recruited from emergency and inpatient acute care. To accomplish these aims, the project will enhance the Opioid Addiction Recovery Support (OARS), an existing Q2i company technology, with a new evidence-based reward, contingency management (CM) function. CM interventions systematically reward (reinforce) specific behaviors like treatment initiation and adherence with therapy attendance and drug-free urine tests and are highly efficacious. An OARS solution enhanced with a CM component (OARSCM) that allows for the automatic calculation, delivery, and redemption of rewards contingent on objective evidence of treatment behaviors may be key to improving Suboxone initiation and adherence. In Phase 1 of this proposal, the existing OARS clinician portal and patient mobile application will be modified to accommodate entry into the software system from an acute care setting and to automatically manage and deliver rewards to create OARSCM using patient-centered design principles. Focus groups with OUD patients and other key stakeholders will inform design. Primary usability outcomes will be examined, and the program iteratively updated. After meeting milestones, there was a proof-of-concept pilot of usability, acceptability, and effects on initial behavior targets with approximately 20 patients and at least 4 providers.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. Presenting for acute care at UMass University and Memorial hospitals, including EDs, inpatient medical units, or inpatient behavioral health units for opioid addiction related health complaints, including opioid overdose, opioid related medical consequences, opioid intoxication or withdrawal syndromes, and/or seeking help for OUD
3. Presence of a current DSM-V opioid use disorder (OUD), mild to severe
4. Medically appropriate for outpatient Suboxone treatment, as judged by the treating clinician and behavioral health consultant or toxicologist working with the patient clinically

Exclusion Criteria:

1. Persistent altered mental status (not alert, not oriented, psychotic).
2. Not interested or willing to participate in Suboxone treatment
3. Best referral site is NOT one of the study's partner clinics in the central MA region, which will be outpatient MAT clinics and primary care within the UMass system and the three other primary facilities outside of the UMass system.
4. Unwilling to use the OARSCM app (if assigned)
5. Does not have access to their own smartphone with at least iOS 7.1 or Android 4.2, the minimal technology required to run the app, or not willing to access clinic-dedicated computer to access the program
6. Currently in state custody or pending legal action that might lead to imprisonment
7. Cannot paraphrase the study requirements
8. Does not read or speak English
9. Does not reside in the central MA region
10. Already enrolled in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Davis-Martin, PhD, Study Director — University of Massachusetts Chan Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all individual participant data (IPD) that underlie published results.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available starting 6 months after publication of results.
Access Criteria: Deidentified data will be accessible to researchers who wish to conduct analyses not reported in prior publications. The study principal investigator will review any request for data to ensure no overlapping analyses. Deidentified data will be shared via secure, HIPAA-compliant data transfers.

REFERENCES:
- See also: Webpage for OARSCM solution — https://q2i.com/oars-cm/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Usability testing participants: Patients: n=12, Providers: n=4; Proof-of-concept field test participants: Patients: n = 11
  (1 patient participated in both usability and field test portions of the study, overall study N = 26)
Groups:
- OARSCM Patients: After successful completion of usability testing (Patients: n=12, Providers: n=4), a proof-of-concept field test was completed. OARSCM patients (n = 10) received TAU procedures during enrollment (SBIRT for opioid use disorder and a warm handoff to outpatient MOUD treatment). TAU outpatient MOUD treatment consists of urine toxicology (Utox) screening, group/individual therapy, and MOUD prescription. Treatment visits are typically weekly in weeks 1-4 and taper over time. Patients earned chances for prizes, for targeted behaviors, which escalated for each targeted behavior in a row, with reset criteria. For scheduling a MOUD treatment intake, patients will earn 2 chances for prizes. Chances for prizes will increase by 2 chances with each targeted behavior in a row up to a max of 10 draws/targeted behavior. There are 18 targeted behaviors during the 4-week field test (schedule intake, complete intake, 4 opioid-negative Utox/week plus bonuses for cocaine-negative Utox, and 4 therapy/week).
  Software Application: Access is granted to participants for 4 weeks to the OARSCM platform which includes reinforcements for meeting MOUD treatment goals.
- Usability Testing Patients; Usability Testing Providers: After successful completion of usability testing (Patients: n=12, Providers: n=4), a proof-of-concept field test was completed. OARSCM patients (n = 10) received TAU procedures during enrollment (SBIRT for opioid use disorder and a warm handoff to outpatient MOUD treatment). TAU outpatient MOUD treatment consists of urine toxicology (Utox) screening, group/individual therapy, and MOUD prescription. Treatment visits are typically weekly in weeks 1-4 and taper over time. Patients earned chances for prizes, for targeted behaviors, which escalated for each targeted behavior in a row, with reset criteria. For scheduling a MOUD treatment intake, patients will earn 2 chances for prizes. Chances for prizes will increase by 2 chances with each targeted behavior in a row up to a max of 10 draws/targeted behavior. There are 18 targeted behaviors during the 4-week field test (schedule intake, complete intake, 4 opioid-negative Utox/week plus bonuses for cocaine-negative Utox, and 4 therapy/week).
Period: Usability Testing (1 Day)
Arm/Group | OARSCM Patients | Usability Testing Patients | Usability Testing Providers
Started | 0 | 12 | 4
Completed | 0 | 12 | 4
Not Completed | 0 | 0 | 0
Period: Field Testing (4 Weeks)
Arm/Group | OARSCM Patients | Usability Testing Patients | Usability Testing Providers
Started | 11 | 0 | 0
Completed | 10 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Usability testing participants: Patients: n=12, Providers: n=4; Proof-of-concept field test participants: Patients: n = 11
  (1 patient participated in both usability and field test portions of study, reported here in the OARSCM Patients section)
Groups:
- OARSCM Patients: After successful completion of usability testing (Patients: n=12, Providers: n=4), a proof-of-concept field test was completed. OARSCM patients (n = 10) received TAU procedures during enrollment (SBIRT for opioid use disorder and a warm handoff to outpatient MOUD treatment). TAU outpatient MOUD treatment consists of urine toxicology (Utox) screening, group/individual therapy, and MOUD prescription. Treatment visits are typically weekly in weeks 1-4 and taper over time. Patients earned chances for prizes, for targeted behaviors, which escalated for each targeted behavior in a row, with reset criteria. For scheduling a MOUD treatment intake, patients will earn 2 chances for prizes. Chances for prizes will increase by 2 chances with each targeted behavior in a row up to a max of 10 draws/targeted behavior. There are 18 targeted behaviors during the 4-week field test (schedule intake, complete intake, 4 opioid-negative Utox/week plus bonuses for cocaine-negative Utox, and 4 therapy/week).
  Software Application: Access is granted to participants for 4 weeks to the OARSCM platform which includes reinforcements for meeting MOUD treatment goals.
  *1 participant completed both OARSCM Patient arm and Usability Patient arm (listed only under OARSCM Patient arm here)
- Usability Patients: After successful completion of usability testing (Patients: n=12, Providers: n=4), a proof-of-concept field test was completed. OARSCM patients (n = 10) received TAU procedures during enrollment (SBIRT for opioid use disorder and a warm handoff to outpatient MOUD treatment). TAU outpatient MOUD treatment consists of urine toxicology (Utox) screening, group/individual therapy, and MOUD prescription. Treatment visits are typically weekly in weeks 1-4 and taper over time. Patients earned chances for prizes, for targeted behaviors, which escalated for each targeted behavior in a row, with reset criteria. For scheduling a MOUD treatment intake, patients will earn 2 chances for prizes. Chances for prizes will increase by 2 chances with each targeted behavior in a row up to a max of 10 draws/targeted behavior. There are 18 targeted behaviors during the 4-week field test (schedule intake, complete intake, 4 opioid-negative Utox/week plus bonuses for cocaine-negative Utox, and 4 therapy/week).
  *1 participant completed both OARSCM Patient arm and Usability Patient arm (listed only under OARSCM Patient arm here)
- Usability Providers: After successful completion of usability testing (Patients: n=12, Providers: n=4), a proof-of-concept field test was completed. OARSCM patients (n = 10) received TAU procedures during enrollment (SBIRT for opioid use disorder and a warm handoff to outpatient MOUD treatment). TAU outpatient MOUD treatment consists of urine toxicology (Utox) screening, group/individual therapy, and MOUD prescription. Treatment visits are typically weekly in weeks 1-4 and taper over time. Patients earned chances for prizes, for targeted behaviors, which escalated for each targeted behavior in a row, with reset criteria. For scheduling a MOUD treatment intake, patients will earn 2 chances for prizes. Chances for prizes will increase by 2 chances with each targeted behavior in a row up to a max of 10 draws/targeted behavior. There are 18 targeted behaviors during the 4-week field test (schedule intake, complete intake, 4 opioid-negative Utox/week plus bonuses for cocaine-negative Utox, and 4 therapy/week).
- Total: Total of all reporting groups
Arm/Group | OARSCM Patients | Usability Patients | Usability Providers | Total
Number analyzed (Participants) | 11 | 11 | 4 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (8.99) | 32 (10.11) | 35 (5.57) | 33 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 3 | 9
  Male | 10 | 6 | 1 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 9 | 11 | 4 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 9 | 10 | 3 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 4 | 26

OUTCOME MEASURES:

1. Primary Outcome: OARSCM Usability - Phase 1 Usability
Description: ≥ 3 participants in a row use the program without staff assistance and no more substantive improvements are needed
Time Frame: during usability sessions with participants at the time of study enrollment, 1 day
Measure: Count of Participants; unit: Participants
Groups:
- OARSCM Usability Testing: Participants completed Usability and Acceptability Testing.
Arm/Group | OARSCM Usability Testing
Number analyzed (Participants) | 12
Participants | 12

2. Primary Outcome: OARSCM Acceptability - Phase 1 Usability
Description: Acceptability outcome will be an average System Usability Scale score of ≥ 80 (range 0-100), with higher numbers indicative of better scores
Time Frame: during usability sessions with participants at the time of study enrollment, 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- OARSCM Usability Testing: Participants completed the System Usability Scale (scores range 0-100), with higher numbers indicative of better scores.
Arm/Group | OARSCM Usability Testing
Number analyzed (Participants) | 12
score on a scale | 93.2 (7.99)

3. Primary Outcome: OARSCM Usability - Phase 1 Field Test
Description: ≥ 3 participants in a row use the program without staff assistance and no more substantive improvements are needed
Time Frame: End of 4-week field test period
Measure: Count of Participants; unit: Participants
Groups:
- OARSCM Field Testing: After successful completion of usability testing (Patients: n=12, Providers: n=4), a proof-of-concept field test was completed. OARSCM patients (n = 11) received TAU procedures during enrollment (SBIRT for opioid use disorder and a warm handoff to outpatient MOUD treatment). TAU outpatient MOUD treatment consists of urine toxicology (Utox) screening, group/individual therapy, and MOUD prescription. Treatment visits are typically weekly in weeks 1-4 and taper over time. Patients earned chances for prizes, for targeted behaviors, which escalated for each targeted behavior in a row, with reset criteria. For scheduling a MOUD treatment intake, patients will earn 2 chances for prizes. Chances for prizes will increase by 2 chances with each targeted behavior in a row up to a max of 10 draws/targeted behavior. There are 18 targeted behaviors during the 4-week field test (schedule intake, complete intake, 4 opioid-negative Utox/week plus bonuses for cocaine-negative Utox, and 4 therapy/week).
  Software Application: Access is granted to participants for 4 weeks to the OARSCM platform which includes reinforcements for meeting MOUD treatment goals.
Arm/Group | OARSCM Field Testing
Number analyzed (Participants) | 11
Participants | 11

4. Primary Outcome: OARSCM Acceptability - Phase 1 Field Test
Description: as for outcome 2
Time Frame: End of 4-week field test period
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- OARSCM Field Testing: Participants completed the System Usability Scale (scores range 0-100), with higher numbers indicative of better scores
Arm/Group | OARSCM Field Testing
Number analyzed (Participants) | 8
score on a scale | 78.1 (20.78)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | OARSCM
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT05159362/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT05159362/SAP_001.pdf